CLINICAL TRIAL: NCT06022393
Title: CBT-Training Zur Kognitiven Umbewertung Als Lntervention Bei Patienten*Innen Mit Funktionellem Tremor - Eine EEG-Studie
Brief Title: CBT Training for Cognitive Reappraisal as an Intervention for Patients With Functional Tremor - an EEG Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Graz (Other)
Collaborators: University of Graz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 35-315 ex 22/23
Record Dates: First submitted 2023-07-17; First posted 2023-09-01 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2023-09

CONDITIONS: Functional Movement Disorder
Keywords: EEG; Psychology; neuropsychology; cognitive reappraisal; cognitive behavioral therapy; Emotional Regulation
MeSH Terms: conditions — Conversion Disorder; Emotional Regulation | interventions — Microscopy, Interference

STUDY DESIGN:
Intervention Model Description: The patients are randomly assigned to one of two groups. The intervention group completes CBT-training to improve their cognitive reappraisal and consequently their emotion-regulation-skills and the control group completes tasks that ask them to reflect about their daily lifes.
Who Masked: Participant, Outcomes Assessor
Masking Description: The patients are randomly assigned to a group and do not know whether that is the intervention or the control group.
  The physicians conducting the preliminary assessments do not know which group the patient was placed in.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cognitive Reappraisal (Experimental): The intervention group completes CBT-training to improve their cognitive reappraisal and emotion-regulation-skills.
  Interventions: Behavioral: Cognitive Reappraisal
- Reflection (Sham Comparator): The control group completes tasks based on reflection about their daily lifes, which should have no impact on their emotion-regulation-skills or functional motor disorder.
  Interventions: Behavioral: Reflection

INTERVENTIONS:
Behavioral: Cognitive Reappraisal — Patients complete 14 tasks on an app in a time span of 4 weeks in which they are asked to cognitively reappraise fear or anger inducing situations and are encouraged to implement this strategy into their daily lifes.
  Arms: Cognitive Reappraisal
Behavioral: Reflection — Patients complete 14 tasks on an app in a time span of 4 weeks in which they are asked to reflect on certain topics of their day.
  Arms: Reflection

SUMMARY:
The aim of this psychological study is to evaluate the effect of a cognitive behavioral therapy (CBT) intervention aimed at improving cognitive reappraisal on (1) Clinical and Self-Rated Health according to Patient Global Impression-Change (PGI-C), Patient Global Impression-Severity (PGI-S), Clinical Global Impression-Change (CGI-C) and Clinical Global Impression-Severity (CGI-S) after 4 weeks, (2) the change in the severity of the functional movement disorder/tremor as assessed by a blinded clinician using the Simplified Version of the Psychogenic Movement Disorders Rating Scale (S-FMDRS) after 4 weeks and (3) the change in the severity of functional tremor assessed via the Fahn Tolosa Marin Tremor Rating Scale (FTM) after 4 weeks.

The knowledge gained about the introspective and neurobiological effect of this cognitive behavioral therapy intervention should enable improved therapy options for patients with functional tremor / functional motor disorders in the future.

DETAILED DESCRIPTION:
This is an intervention study including patients of the outpatient clinic for movement disorders at the University Clinic of Neurology in Graz.

The patients will randomly be assigned to the intervention (cognitive reappraisal) or control (reflection) group.

The study consists of a first preliminary examination at the University clinic, followed by an electroencephalogram (EEG)-lab-session at the Institute of Psychology of the Karl-Franzens-University of Graz. The patients will complete emotion-regulation tasks while the EEG is conducted and then be introduced to an App, with which they will either complete 14 cognitive-reappraisal-tasks (intervention) or 14 reflection-tasks (control) within the next 4 weeks. A task will need to be completed in the App once every two days.

After this training period, there will be a second preliminary examination at the University Clinic as well as a second subsequent EEG-lab-sessions at the Institute of Psychology at the Karl-Franzens-University.

In addition, after two weeks of training, the patients will receive a short phone call and will be asked to complete the PGI-S and PGI-C.

Questionnaires completed during the first preliminary examination:

1. CGI-S - Clinical Global Impression - severity
2. PGI-S - Patient Global Impression - severity
3. FTM - Fahn Tolosa Marin Tremor Rating Scale
4. S-FMDRS - Simplified Version of the Psychogenic Movement Disorders Rating Scale

Questionnaires completed during the first EEG-lab-session:

1. VKT - Verbal creativity test
2. RIT - Reappraisal Inventiveness Test
3. ERQ - Emotion Regulation Questionnaire
4. LPFS-BF - Level of Personality Functioning Scale:
5. SF-36 - Short Form (36)
6. EQ-5D-5L - Health Questionnaire
7. PAHD - Psychosomatic Assessment Health-DISC

Questionnaires completed during the second preliminary examination:

All the questionnaires also used in the first examination plus:

1. CGI-C - Clinical Global Impression - Change
2. PGI-C - Patient Global Impression - Change

Questionnaires completed during the second EEG-lab-session:

The same as in the first EEG-lab-session.

4 weeks after the completion of the last EEG-lab-session, the patients will receive another short phone-call in which they will again be asked to complete the PGI-S and PGI-C.

ELIGIBILITY:
Inclusion Criteria:

- Diagnosis of a functional movement disorder

Exclusion Criteria:

* The patient is not capable of giving consent.
* The patient does not have sufficient knowledge of German to answer the questionnaires (questionnaires are only available in German).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-08-16 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2025-08-31 (Actual)

PRIMARY OUTCOMES:
Change in Clinical health - Clinical Global Impression Severity Scale | 4 weeks
  Clinical health according to Clinical Global Impression of Severity Scale (CGI-S) rated by a medical professional.
  Three questions regarding patients current mood, influence of the symptoms on everyday motor function and overall severity.
  Answer options:
  1. Not at all/very easy
  2. Lightly
  3. Moderate
  4. Strong
  5. Very strong Higher values = worse outcome
Change in Clinical health - Clinical Global Impression of Change | 4 weeks
  Clinical health according to Clinical Global Impression of Change Scale (CGI-C) rated by a medical professional.
  Three questions regarding patients mood, everyday motor function and overall change as well as a rating regarding the relevance of the change (Yes or No). Answer options:
  Very Much worse Much worse Slightly worse No change Marginally better Much better Very Much better
  Higher values = better outcome
Change in Self-assessed health - Patient Global Impression Severity Scale | 4 weeks
  Self-assessed health according to Patient Global Impression of Severity Scale (PGI-S) rated by the patients themselves.
  Three questions regarding patients current mood, influence of the symptoms on everyday bodily function and overall severity.
  Answer options:
  1. Not at all/very easy
  2. Lightly
  3. Moderate
  4. Strong
  5. Very strong Higher values = worse outcome
Change in Self-assessed health - Patient Global Impression of Change | 4 weeks
  Self-assessed health according to Patient Gloabal Impression of Change Scale (PGI-C) rated by the patients themselves.
  Three questions regarding patients mood, everyday bodily function and overall change as well as a rating regarding the relevance of the change (Yes or No). Answer options:
  Very Much worse Much worse Slightly worse No change Marginally better Much better Very Much better
  Higher values = better outcome
The change in severity of the functional movement disorder | 4 weeks
  The change in severity as assessed by a blinded clinician using the severity of the functional movement disorder by means of the Simplified Version of the Psychogenic Movement Disorders Rating Scale (S-FMDRS). Scoring: 0-3, higher values indicate worse outcome.
The change in tremor severity | 4 weeks
  The change in tremor severity assessed using the Fahn Tolosa Marin Tremor-Rating-Scale.
  Scoring: 0-4, higher values indicate worse outcome.

SECONDARY OUTCOMES:
Change in the ability of emotion regulation | 4 weeks
  The change in the ability of emotion regulation assessed using the Emotion Regulation Questionnaire.
  High scores on the reassessment scale suggest that the person is more likely to use cognitive strategies to change the emotional meaning of situations. This may be associated with better emotional adaptability and well-being.
  High scores on the suppression scale indicate that the person is more inclined to suppress or avoid the expression of emotions. This may be associated with lower emotional adaptability and well-being.
Changes in patients EEG-activity. | 4 weeks
  Training-based changes in patients' EEG activity will be assessed for a) tasks-related changes in EEG alpha frequency power (TRPs) as well as b) frontal alpha asymmetry changes during the generation of cognitive reappraisals. Changes in these parameters should unterline behavioral changes in reappraisal success, divergent thinking, and executive functioning. Moreover, we will look at c) the EEG theta/beta frequency ratio to map changes in stress coping, emotion regulation, and behavioral flexibility.
Change in the patients Creativity | 4 weeks
  The change in creativity assessed using the Verbal Creativity Test. No Minimum or Maximum values, higher score = better outcome.
Change in the patients Welfare- Health Questionnaire EQ-5D-5L. | 4 weeks
  The change in the patients welfare assessed using the Health Questionnaire EQ-5D-5L.
  5 Level, Scores: 1-5, higher values indicate worse outcome.
  1 overall Scale: 0-100, higher values indicate better outcome.
Change in the patients Welfare- Short Form Health Questionnaire | 4 weeks
  The change in the patients welfare assessed using the Short Form Health Questionnaire.
  The possible score ranges from 0 to 100 points, with 0 points representing the greatest possible restriction of health, while 100 points indicate no health restriction.
Change in the patients Welfare - Psychosomatic Assessment Health-DISC. Minimum value in each section: 0 Maximum value in each section: 10 Higher scores = better outcome. | 4 weeks
  The change in the patients welfare assessed using the Psychosomatic Assessment Health-DISC 6 Levels, Scores: 0-10, higher values indicate better outcome.
Change in patients personality and behavioral aspects | 4 weeks
  The change in patients personality and behavioral aspects assessed using the Level of Personality Functioning Scale.
  The items are on a 4-point Likert scale from 1 ("doesn't apply at all") to 4 ("applies exactly") to"). The evaluation is carried out by means of summaries, so that values on the Overall scale: 12 - 48 Subscales Self and Interpersonal: 6 - 24
Long-term change in Self-assessed health - Patient Global Impression of Change | 8 weeks
  Self-assessed health according to Patient Global Impression of Change Scale (PGI-C) rated by the patients themselves.
  Three questions regarding patients mood, everyday bodily function and overall change as well as a rating regarding the relevance of the change (Yes or No). Answer options:
  Very Much worse Much worse Slightly worse No change Marginally better Much better Very Much better Higher values = better outcome
Long-term change in Self-assessed health - Patient Global Impression Severity Scale | 8 weeks
  Self-assessed health according to Patient Global Impression of Severity Scale (PGI-S) rated by the patients themselves.
  Three questions regarding patients current mood, influence of the symptoms on everyday bodily function and overall severity.
  Answer options:
  1. Not at all/very easy
  2. Lightly
  3. Moderate
  4. Strong
  5. Very strong Higher values = worse outcome

CONTACTS AND LOCATIONS:
Overall Officials: Corinna Perchtold-Stefan, PhD, Study Chair — University of Graz; Petra Schwingenschuh, MD, Study Chair — Medical University of Graz
Locations (1):
- Medical University of graz, Graz, Styria, Austria

IPD SHARING:
Plan to Share IPD: No